CLINICAL TRIAL: NCT03152851
Title: The Effect of Sonographic Bladder Compressive Stimulation Technique for Bag Urine Collection in Pediatrics: Randomized Controlled Trial
Brief Title: The Effect of Sonographic Bladder Compressive Technique for Bag Urine Collection in Pediatrics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyuksool Kwon, Clinical assistant Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: B-1609-362-001
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure stimulus group by ultrasound probe (Experimental): A pressure stimulus would be applied once using a device (ultrasound probe) to the anteroposterior wall of the bladder until the anterior & posterior wall meet if the measured diameters (AP x T) is 2 X 2 or more by ultrasound
  Interventions: Procedure: Pressure stimulus group
- Non-pressure stimulus group (No Intervention): No pressure stimulus would be given

INTERVENTIONS:
Procedure: Pressure stimulus group
  Arms: Pressure stimulus group by ultrasound probe

SUMMARY:
Aim: to shorten the time of urination by bladder pressure stimulation in children less than 36 months of age who need urinalysis to exclude or diagnose urinary tract infections and to speed up the start time of antibiotics treatment or to eliminate the overcrowding of emergency room(ER) by shortening the time of ER stay.

DETAILED DESCRIPTION:
* According to preassigned 1:1 randomization of 40 patients assigend to intervention group and other 40 patients assign to control group as follow.
* Get documented agreement from the caregiver if the patient meets the criteria.
* While the a nurse attaches a kismo to a patient, the researcher at the bedside measures the patient's bladder size as an maximal anteroposterior (AP) and transverse (T) diameter(cm)
* If the measured diameters (AP x T) is 2 X 2 or more, the research assistant check the assigned group of the patient.
* If the patient assigned to the intervention group, a pressure stimulus is applied once using an ultrasonic probe to the anteroposterior wall of the bladder until the anterior & posterior wall meet.
* If the AP X T was less than 2 X 2, excluded from the study enrollment.
* During the study, caregivers and the assigned nurse will be blinded

ELIGIBILITY:
Inclusion Criteria:

* Body temperature of patients ≥ 38℃ reported by guardians
* No definite focus of fever detected by physical examination
* Guardian agrees to use urine bag(kismo) collection technique

Exclusion Criteria:

* Previous history of urinary tract infections
* Underlying urinary tract diseases (eg congenital anomalies, neuroblastomas, already diagnosed bladder ureters)
* ICU treatment indicated
* Newly diagnosed hydronephrosis on the day of visit

Ages: 3 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
The urine collection time | up to 2 hours
  The urine collection time

SECONDARY OUTCOMES:
The antibiotic administration time | up to 1 day
  The antibiotic administration time
Emergency department(ED) length of stay time | up to 1 day
  Emergency department(ED) length of stay time
Comparison between the patients who were diagnosed as actual urinary tract infections and those who were not. | up to 1 day
  Comparison between the patients who were diagnosed as actual urinary tract
Complications | up to 1 month
  Complications

CONTACTS AND LOCATIONS:
Overall Officials: JAEYOON JUNG, MD PhD, Principal Investigator — The Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - The Seoul National Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoum national university, Seoul

IPD SHARING:
Plan to Share IPD: Undecided